CLINICAL TRIAL: NCT05648266
Title: Serratus Plane Block After Minimally Invasive Mitral Valve Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 19518181202119
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Minimal Invasive Cardiac Surgery; Minimal Invasive Cardiac Surgery Mitral Valve Surgery; Serratus Anterior Plane Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous SAPB (Active Comparator): postoperative serratus-anterior-plane-block 20ml Ropivacain 0,75%, pain catheter with continous administered Ropivacain (5ml/h 0,2% for 48h)
  Interventions: Drug: Continous SAPB (Ropivacain); Other: institutional standard of care pain medication protocol
- Placebo (Placebo Comparator): standard of care
  Interventions: Other: institutional standard of care pain medication protocol

INTERVENTIONS:
Drug: Continous SAPB (Ropivacain) — postoperative SAPB and pain catheter with continous administered (5ml/h Ropivacain 0,2%) for 48h
  Arms: Continuous SAPB
Other: institutional standard of care pain medication protocol — institutional standard of care pain medication protocol

SUMMARY:
Patients undergoing minimally invasive mitral valve reconstruction via small thoracotomy are randomized into two groups.

The intervention group receives serratus anterior plane block after minimally invasive mitral-valve reconstruction, following 48h infusion with ropivacaine 2% continually.

The control group receives a placebo pump without infusion. Primary endpoints are perceived pain using a numeric pain rating scale and opioid consumption during the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

-Planned minimal invasive mitral valve repair via right anterior thoracotomy

Exclusion Criteria:

* Pregenancy
* Opioid abuse
* Historyof chronic pain
* Allergy to local anaesthetics (in this case ropivacain)
* Patients who simultaneously participate in another interventional clinical trial, unless the Principal Investigators of the clinical trials give consent by mutual agreement Soft tissue infection in the area of the procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Difference of Numeric Rating Scale after MIC-MKR | within 12, 24 and 48 hours after surgery
  Numeric Rating Scale (0-10, 0=smallest value, 10=greatest value)

SECONDARY OUTCOMES:
Difference of opioid consumption after MIC-MVR | within 12, 24 and 48 hours after surgery
  daily, cumulative dose of opioid analgetic medication after MIC-MKR

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hamburg Eppendorf, Hamburg, Hamburg, Germany